CLINICAL TRIAL: NCT04688840
Title: Smartphone Application: A Possible Solution for Follow up of Patients With Hip Arthroplasty During COVID-19 Pandemic
Brief Title: Smartphone Application: A Possible Solution for Follow up of Patients With Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, ahmed m. samy, assisstant professor, Tanta University
Other Study IDs: TantaH
Record Dates: First submitted 2020-12-14; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Telemedicine
Keywords: Whatsapt; hip arthroplasty; Telemedicine; patient's satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study results and satisfaction with telemedicine: the investigators designed a group on WhatsApp for all patients included in the study. The questionnaires were sent on the group to be filled by the patients in addition to a request for routine x ray follow up. Also, the investigators used the group to send any announcement, schedule of routine visits and some instructions about how to answer the questionnaires. To keep the privacy of patients' informations, every patient was asked to resend the file and x- ray pictures to the surgeon private account. the investigators collected data received by all patients and reviewed all x-rays. If there was any serious complain or major radiological finding the investigators asked the patient for immediate clinical visit.
  Interventions: Procedure: hip arthropalsty
- study results and satisfaction with routine follow up: the investigators asked the patients to come for routine follow up visit (RV) and reevaluate them clinically and radiologically. the investigators asked patients to calculate total time needed for completion of the questionnaires, time needed for x-ray and the investigators added time needed for reviewing these files. The same was done at the RV including time of transportation
  Interventions: Procedure: hip arthropalsty

INTERVENTIONS:
Procedure: hip arthropalsty — follow up of patients with primary hip arthroplasty with at least one year follow up electronically and by routine method

SUMMARY:
Introduction: Over the last decades, telemedicine has been used in many surgical aspects. Its role in postoperative follow up is of significant interest with a remarkable success. Since the appearance of COVID-19, the challenge is how to follow the recommendations of World Health Organization which stressed on the importance of social distancing to avoid infection and at the same time provides satisfactory medical services. This study was done to evaluate the feasibility and efficacy of Whatsapp social media program in postoperative follow up of patients with primary hip arthroplasty at the time of pandemic

DETAILED DESCRIPTION:
This is a prospective randomized comparative study. The investigators reviewed all registered patients underwent primary total hip arthroplasty (T.H.A.) at our department up to five years ago. Four hundred sixty three patients were recorded at our data base. After reviewing patients' files, the investigators excluded fifty two patients with follow up less than one year and 29 patients with a previous history of complications. Three hundred eighty two patients were initially eligible for the study. The investigators contacted them by telephone calls in order to ask them to be included in this study. The investigators were unable to contact 57 patients, 51 refused to be included, 31 preferred a personal contact with the surgeon, 14 patients were died and 51 patients did not have an internet access. One hundred seventy eight participants were finally eligible to be included in our research. Only 167 participants completed both electronic and routine follow up and these were our final materials. The investigators designed a group on WhatsApp for all participants included in the study. The questionnaires were sent on the group to be filled by the participants in addition to a request for routine x ray follow up. Also, the investigators used the group to send any announcement, schedule of routine visits and some instructions about how to answer the questionnaires. To keep the privacy of participants' information, every one was asked to resend the file and x- ray pictures to the surgeon private account. The investigators collected data received by all participants and reviewed them. If there was any serious complain or major radiological finding the investigators asked the participant for immediate clinical visit. One month later, the investigators started to recall all participants for routine follow up visit (RV) and reevaluate them clinically and radiologically. The investigators asked participants to calculate total time needed for completion of the questionnaires, time needed for x-ray and we added time needed for reviewing these files. The same was done at the RV including time of transportation. The investigators obtained a written consent from all of the participants after discussion about the aim of the research and the confidentiality of their data. All procedures performed in the study were in accordance with the ethical standards of our department and with the 1964 Helsinki declaration and its later amendments.

the investigators evaluated the effectiveness of the electronic visit (EV) by calculation of the number of missing complications or signs detected at the time of RV and require any interference or close observation

ELIGIBILITY:
inclusion criteria:

* patients underwent primary hip arthroplasty for at least one year ago
* familiarity of the patient or one of close relative (e.g. son or daughter) with smart phone applications.

Exclusion Criteria:

* patients that have no facility or experience with computer or internet and do not have a close relative to assist them
* patients with any previous complications (e.g. Infection, dislocation and loosening).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with primary total hip arthroplasty without history of postoperative complications
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) | 7 months
  evaluate the function ad activity of the hip joint
Short Form Health Survey Clinical care (SF12) | 7 months
  describe general health status of the participant
Self-Administered Patient Satisfaction Scale (SAPS) | 7 months
  satisfaction of the participants with the method of follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Samy, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
when i publish the data